CLINICAL TRIAL: NCT04874623
Title: Identification of IgA Monoclonal Antibodies Anti-Clostridium Difficile Surface Proteins
Brief Title: Monoclonal Antibodies in Clostridium Difficile Infection
Acronym: IgAClostridium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP180354
Record Dates: First submitted 2020-09-22; First posted 2021-05-06 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Clostridium Infection
Keywords: Clostridium difficile infection; Therapeutic monoclonal antibodies
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDI (Experimental)
  Interventions: Other: Collection of peripheral blood mononuclear cells

INTERVENTIONS:
Other: Collection of peripheral blood mononuclear cells — Analysis of specific memory B cells in CDI patients

SUMMARY:
Immunoglobulin A (IgA), the major mucosal antibody, plays a key role in maintaining diversity of the intestinal microbiota and eliminating intestinal pathogens. Dysbiosis is an important risk factor for Clostridium difficile infection, which is the leading cause of nosocomial diarrhea in industrialized countries. This study aims to develop IgA monoclonal antibodies targeting C. difficile surface proteins.

DETAILED DESCRIPTION:
Immunoglobulin A (IgA), the major mucosal antibody, plays a key role in maintaining the diversity of the intestinal microbiota and eliminating intestinal pathogens. They modulate microbiota composition and also commensal bacteria homeostasis, thus promoting a symbiotic relationship. These observations, derived from mouse studies, open promising therapeutic perspectives: IgA could be used to restore or maintain a healthy microbiota in individuals suffering from intestinal dysbiosis. Specific to a pathogen, IgA can also be considered as an alternative to antibiotics by mimicking a physiological elimination.

Abnormalities in microbial diversity (i.e. dysbiosis) have been associated in humans with various diseases such as Clostridium difficile infection, which is the leading cause of nosocomial diarrhea in industrialized countries. The incidence of CDI has dramatically raised since the early 2000s, with an increasing severity. Current treatments are limited to the administration of antibiotics that unbalance the intestinal microbiota, a risk factor for relapse. These frequent relapses contribute to the severity and chronicity of the infection.

This study aims to generate human IgA-type antibodies targeting C. difficile surface proteins with neutralizing and/or protective activity. These antibodies will be selected against surface proteins involved in the early stages of colonization. After injection or ingestion, these IgA antibodies should reproduce physiological mucosal immunity, treat severe forms and prevent the occurrence of C. difficile relapses while limiting deleterious effects on the intestinal microbiota.

C. difficile-specific B cells will be selected from infected patients. After selection of the most neutralizing IgA antibodies in vitro, these will be administered to C. difficile infected mice.

ELIGIBILITY:
Inclusion Criteria:

* adult patient, 18 years of age
* diarrhea and/or abdominal pain.
* Presence of C. difficile toxins in feces
* Patient having dated and signed informed consent.

Exclusion Criteria:

* pregnant or nursing women
* adult under guardianship
* Ileus
* Peritonitis
* Pseudomembranous colitis
* Hemodynamic instability
* Fever ≥ 38.5°C
* Shivers
* Respiratory failure
* Leukocytosis > 15x109/L
* Serum creatinin >50% reference values)
* Serum lactate > 5mM
* Serum Albumine < 30g/l
* Other diarrhea cause
* Humoral immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Generate C. difficile specific antibodies from circulating memory B lymphocytes of C. difficile patients. | From the blood samples taken between Day 1 and Day 7 after the diagnostic of CDI
  The presence of SlpA and Cwp84 specific memory B cells will be assessed from a single sample per patient. After separation of blood mononuclear cells, specific memory B cells will be selected using microfluidic drop technology. The variable VH and VL fragments of the immunoglobulins, which define the specificity of the antibodies, will be sequenced for each selected B cell. The corresponding antibodies will then be produced in a well-established cell line.

SECONDARY OUTCOMES:
Antibody affinity assessment | From the blood samples taken between Day1 and Day7 after the diagnostic of CDI
  The affinity of the antibodies will be evaluated by surface plasmon resonance (Biacore®).
Neutralizing capacity evaluation affinity | From the blood samples taken between Day1 and Day7 after the diagnostic of CDI
  The neutralizing activity will be evaluated in vitro: the capacity of the antibodies to decrease the proliferation of the bacteria (in liquid culture), to decrease its mobility (solid culture), to inhibit biofilm formation and to inhibit its adhesion to the surface of intestinal epithelial cells (quantified using the Caco-213 line).

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste Hervier, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Maladies infectieuses et tropicales, Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No